CLINICAL TRIAL: NCT00248365
Title: Safety, Biological and Clinical Efficacy of Two Intensity Levels of Theralux Extracorporeal Photochemotherapy in Subjects With Extensive Chronic GvHD Refractory or Intolerant to Standard Therapy: A Randomized, Open-label Phase I/II Clinical Trial
Brief Title: Theralux Extracorporeal Photochemotherapy (ECP) in Patients With Extensive Chronic Graft Versus Host Disease (GvHD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kiadis Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-ECP-001
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Graft vs Host Disease
Keywords: Chronic GvHD; Extensive chronic GvHD; Resistant chronic GvHD
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

ARMS (2):
- Low PDT intensity level (Experimental): Theralux extracorporeal photochemotherapy PDT dose: TH9402 0.33μM
  Interventions: Biological: Theralux extracorporeal photochemotherapy
- High PDT intensity level (Experimental): Theralux extracorporeal photochemotherapy PDT dose: TH9402 1.32μM
  Interventions: Biological: Theralux extracorporeal photochemotherapy

INTERVENTIONS:
Biological: Theralux extracorporeal photochemotherapy

SUMMARY:
The purpose of this study is to assess the tolerability and safety of two intensity levels of Theralux extracorporeal photochemotherapy in the treatment of subjects with steroid refractory or intolerant GvHD.

The current hypothesis is that apoptotic cells re-injected into patients induce an immunomodulation effect alleviating the GvHD symptoms. Using the Theralux procedure, the dose of photodynamic treatment may be modulated to achieve the maximal immunomodulatory effects in the treated patients.

The intervention is iterative extracorporeal photochemotherapy of autologous peripheral blood mononuclear cells (PBMC) with a rhodamine-derivative TH9402 (drug) and Theralux (device).

DETAILED DESCRIPTION:
Graft versus host disease (GvHD) remains a major cause of morbidity and mortality related to allogeneic stem cell transplantation. While improvements in immuno-suppressive regimens have reduced the frequency and severity of acute GvHD, the incidence of chronic GvHD (cGvHD) remains unchanged ranging from 30% after sibling matched related donor transplants to over 70% after unrelated donor bone marrow or peripheral blood stem cell transplant. Factors associated with cGvHD include increased donor and recipient age, prior acute GvHD, and the use of alloimmune female donors. Conventional therapeutic approaches for cGvHD, including corticosteroids and immunosuppressive agents, have demonstrated limited efficacy in patients with extensive disease and are associated with high toxicity.

Iterative extracorporeal photopheresis has demonstrated clinical and immunomodulatory activity in subjects with acute and chronic GvHD. The currently available process of ECP has not been controlled for cell number, exposure time, or specific cell populations targeted due to the nature of the procedure. Using the Theralux procedure, defined populations of cells may be targeted, and the intensity of photoactivating agent and exposure can be modulated to achieve the maximal immunomodulatory effects in the treated subjects. This study will attempt to explore the effects of the Theralux procedure under two defined conditions. Response and toxicity will be determined at each intensity level and the dose associated with clinical response and immunomodulatory effects on DC and NK cell populations will be defined as the optimal intensity level for subsequent larger trials.

ELIGIBILITY:
Inclusion Criteria:

* Clinical features compatible with extensive chronic GvHD
* Refractory or intolerant to standard therapy

Exclusion Criteria:

* Pregnant or lactating women
* Underlying concurrent medical condition which would hinder the ability to safely administer the treatment
* Known hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Participation to another investigational trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Signs of toxicity
Chronic GvHD grading
Dose of immunosuppressive medications

SECONDARY OUTCOMES:
ECOG Performance
Survival
Immunomodulatory and Biological effects

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - B.C. Cancer Research Center, Vancouver, British Columbia
  - McMaster University Medical Center, Hamilton, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec

REFERENCES:
- See also: Kiadis Pharma Web page — http://www.kiadispharma.com